CLINICAL TRIAL: NCT05662969
Title: Machine-perfusion for Liver Transplantation in High Versus Low/Mid-volume Centres: an International Multicentre Survey
Brief Title: Machine Perfusion in High vs Low/Mid-volume Liver Transplant Centers: a Multicentre Survey
Acronym: MP-LTx
Status: Completed | Type: Observational
Sponsor: Roberta Angelico (Other)
Responsible Party: Sponsor-Investigator, Roberta Angelico, Principal investigator, Professor, MD, PhD, FEBS, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Other Study IDs: MPLTPTV1
Record Dates: First submitted 2022-11-29; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Organ Preservation Solution
Keywords: machine perfusion; liver transplant; low/mid volume transplant center

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Low/mid-volume liver transplant centres
  Interventions: Device: MACHINE PERFUSION
- High-volume liver transplant centres
  Interventions: Device: MACHINE PERFUSION

INTERVENTIONS:
Device: MACHINE PERFUSION — Different outcomes of MP use in low/mid-volume and high-volume LT centres

SUMMARY:
Introduction: Machine perfusion (MP) was developed to expand the available donor pool and to improve liver transplantation outcomes. Despite optimal results in clinical trials, MP benefit outside of clinical experimentation in unknown. Low/mid volume centres (L/MVCs) may face logistical/economical difficulties that may in turn hamper optimal MP results.

Methods: An Online 22-item survey on the use of machine perfusion for liver transplantation outside of clinical trials, was distributed to worldwide LT centres representatives. Variables of interest included MP logistics, MP technicalities, MP results, post-MP LT results. Responding centres were grouped into high volume centre (HVCs)(defined as >60 LTs per year in 2019) and L/MVCs. Results from HVCs vs L/MVCs were compared.

ELIGIBILITY:
Inclusion Criteria:

* LT centres that use MP
* LT centres which perform LT before pandemic time (before 2019 included)
* LT centres which perform LT from cadaveric donors and living donors

Exclusion Criteria:

* LT centres that not use MP
* LT centres that use MP but on clinical trials

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 67 LT centres divided by a cutoff of 60LT/year in: 31 low/mid-volume LT centres (<60LT/year) and 36 high-volume LT centres (>60 LT/year)
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Liver transplant(LT) centres different use of graft after utilization of machine perfusion (MP) | 12/2021 - 03/2022
  High Volume Centers and Low/Mid Volume centers differ in their rates of graft utilization after Machine perfusion

SECONDARY OUTCOMES:
Liver Transplant outcomes after Machine Perfusion | 12/2021 - 03/2022
  Reported patient survival rates for Liver Transplant after Machine Perfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Roberta Angelico, Rome, Italy